CLINICAL TRIAL: NCT00889148
Title: Multiple Doses of Gabapentin and Postoperative Morphine Consumption in Primary Hip Arthroplasty
Brief Title: Morphine COnsumption in Joint Replacement Patients, With and Without GaBapentin Treatment, a RandomIzed ControlLEd Study
Acronym: MOBILE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Dr. Manyat Nantha-Aree, MD, FRCAT, Hamilton Heath Sciences
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 07-215-THR
Record Dates: First submitted 2009-04-27; First posted 2009-04-28 (Estimated); Last update posted 2011-03-02 (Estimated); Status verified 2009-04

CONDITIONS: Postoperative Pain; Total Hip Replacement
Keywords: hip; arthroplasty; postoperative pain; gabapentin
MeSH Terms: conditions — Pain, Postoperative | interventions — Gabapentin; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gabapentin (Experimental): 600mg of gabapentin will be given orally two hours preoperatively and 200mg for 3 times a day after surgery for three days.
  Interventions: Drug: Gabapentin
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Gabapentin — 600mg gabapentin given 2 hrs preoperatively and 200mg three times a day after surgery for 3 days
  Other Names: Neurontin
  Arms: Gabapentin
Other: Placebo — Half the patients will be randomized to placebo
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
Total hip arthroplasty is amongst the most painful procedures postoperatively, and pain management can be a challenge. Different measures have been introduced to manage severe postoperative pain in these patients. Previous studies have investigated gabapentin in acute postoperative pain and demonstrated reduced postoperative pain, postoperative morphine consumption, morphine related side effects, and postoperative pain scores. To date, this analgesia adjunct has yet to be investigated for total joint arthroplasty patients.

DETAILED DESCRIPTION:
The study was submitted to Health Canada and has received the letter of no objection. A randomized, double-blind, placebo-controlled trial will be conducted. The randomization scheme will be prepared and done by the pharmacy department at McMaster University. Ninety patients undergoing primary hip arthroplasty will be recruited from the preoperative clinic. Forty-five patients in each population will be allocated to a gabapentin group and the other forty-five patients will be allocated to a placebo group.

ELIGIBILITY:
Inclusion Criteria:

* participants aged 19-90
* elective single joint, primary total hip arthroplasty
* use of PCA with morphine for postoperative pain control has been discussed and agreed upon between patient and anesthetist

Exclusion Criteria:

* bilateral total hip arthroplasty
* revision hip arthroplasty
* underlying diseases of epilepsy, seizure, or chronic pain syndrome
* active gastrointestinal bleeding within the last 6 months
* history of non-steroidal anti-inflammatory drug (NSAID) induced asthma
* known or suspected history of drug or alcohol abuse
* participate currently takes gabapentin or pregabalin for any reason
* participant currently takes pain medication that is more potency than codeine or oxycodone (morphine, hydromorphone, meperidine, methadone, fentanyl, including any long acting narcotics)
* known allergy to study medications: gabapentin, morphine, NSAID, acetaminophen
* unable to tolerate morphine
* liver impairments
* kidney impairment or calculated creatinine clearance by Cockcroft-Gault formula is <=60ml/min
* pregnancy or breast-feeding
* participant currently receives associated worker's compensation benefits (WSIB)
* participant unable or unwilling to give written or informed consent
* unable to use PCA

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2007-10; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Amount of morphine consumption | Two years

SECONDARY OUTCOMES:
Side effects | Two years
  Nausea/Vomiting Sedation Pruritis Visual Disturbance Dizziness/Lightheadness
Pain scores | Two years
  Pain score at rest in PACU, POD1, POD2, POD3 Pain score upon passive movement in PACU, POD1, POD2, POD3 Pain score with weighbearing on POD1, POD2, POD3

CONTACTS AND LOCATIONS:
Overall Officials: Manyat Nantha-Aree, MD, Principal Investigator — Hamilton Health Sciences Corporation
Locations (1):
- Hamilton Health Sciences, Hamilton, Ontario, Canada